CLINICAL TRIAL: NCT05304975
Title: BRAIN-Diabetes: Border Region Area Lifestyle Intervention Study for Healthy Neurocognitive Ageing in Diabetes. A Feasibility Randomised Controlled Trial
Brief Title: Border Region Area Lifestyle Intervention Study for Healthy Neurocognitive Ageing Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Western Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Peter Passmore, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 09069PP
Record Dates: First submitted 2022-01-27; First posted 2022-03-31 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Active Comparator): Participants will be provided with written dietary education, meal plan, recipe ideas, tips and suggestions at their baseline and review study visits.
  The exercise intervention will be delivered remotely. Participants will undergo a physical performance assessment at baseline and receive a home exercise resource that has been designed for older adults.
  Cognitive stimulation will be delivered using Brain HQ®, a computer based cognitive training platform, which utilises visuospatial and auditory games to enhance attention, mental processing speed, learning, memory, and low mood.
  Participants will be informed by the research nurse about their blood results, weight and blood pressure and will receive recommendations to visit their GP to change treatment as necessary.
  The 4-month active intervention will be followed by a 2-month self-directed consolidation phase and all participants will be left to their own initiative for a further 3 months
  Interventions: Behavioral: diet; Behavioral: cognitive stimulation; Behavioral: physical activity; Other: risk factor management
- control (Other): this will be routine management of the diabetes condition as per current recommended practice
  Interventions: Other: risk factor management

INTERVENTIONS:
Behavioral: diet — Participants will be provided with written dietary education, meal plan, recipe ideas, tips and suggestions at their baseline visit. Participants will then meet online with the study nutritionist for around 90 minutes for personal dietary advice which will be based on the latest evidence from the MIND (Mediterranean-DASH diet Intervention for Neurodegeneration Delay) diet tailored for the target population. The nutritionist will support participants to set personal dietary goals and to monitor progress in changing towards the MIND diet. If weight loss is indicated, the nutritionist will also advise energy intake to facilitate 5-10% body weight reduction. Following the initial appointment, review meetings with the nutritionist will take place monthly in the first four months, either online or by telephone and lasting up to 60 minutes
  Arms: intervention
Behavioral: cognitive stimulation — Cognitive stimulation will be delivered using Brain HQ® (Posit Science), a computer based cognitive training platform, which utilises games to enhance attention, mental processing speed, learning, memory, and low mood. On 2 occasions during the first month participants will receive a 30-60min training. The aim is to familiarise participants with games and program processes to optimise engagement with the programme.The cognitive training application is available to download on a range of devices. Following training, participants will be asked to log in and complete the training session at least 4 days per week. Each session is expected to last 30 minutes. Individual cognitive training performance will be recorded centrally. Participants will receive feedback of percentage improvement in performance. The program allows remote monitoring of frequency of use and engagement. Therefore, performance, frequency, duration, and type of use will be recorded centrally throughout the study period
  Arms: intervention
Behavioral: physical activity — The exercise intervention will be delivered remotely. Participants will undergo a physical performance assessment at baseline and receive a home exercise written resource that has been designed for older adults and adapted for the current study. It is expected that participants will begin with a basic level of exercise that will increase in frequency and intensity over the first 4 weeks to reach a core required level. In week one, participants will meet online with the trained exercise instructor for around 60 minutes to plan a personalised exercise programme. The instructor will explain the basics of exercise prescription, the foundations of the personal home programme and safety aspects. The instructor will facilitate appropriate exercise goal setting and demonstrate the exercises within the personal programme. Participants will be advised to wear the study pedometer to record their walking activity and complete the exercise diary to record overall step count and daily exercise.
  Arms: intervention
Other: risk factor management — Metabolic and vascular risk factor management. At each study visit (baseline, month 4, month 6 and month 9), participants will be informed by the research nurse about their blood results, weight and blood pressure and will receive recommendations to visit their GP to change treatment as necessary

SUMMARY:
The objective is to evaluate a culturally tailored adaptation of The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER) protocol targeted for individuals with Type 2 diabetes mellitus (DM) living in the border areas of Ireland. The primary research question to be addressed is; what is the feasibility and acceptability of implementing a multicomponent intervention for the target population in a community setting in comparison to standard clinical care. The study protocol was informed by a phase 1 qualitative study (REC ref 19/NI/0011) involving the target population i.e. older people with Type 2 DM from the border areas of N Ireland and the Republic of Ireland and has been amended (version 2.0) in response to the coronavirus pandemic

DETAILED DESCRIPTION:
Dementia is the most frequent neurodegenerative condition and poses a major health burden with high socioeconomic costs. Attempts to find pharmacologic treatments have been largely unsuccessful, prompting a focus on interventions aimed at modifying risk factors for dementia that occur throughout the life course. In terms of risk factors for dementia, strongest support is for depression, (midlife) hypertension, physical inactivity, DM, (midlife) obesity, hyperlipidaemia, and smoking. The incidence of any dementia was approximately two-to three-fold higher in people with than in those without DM, leading to suggestions that interventions addressing lifestyle changes and DM treatment could be beneficial.

A number of intervention studies in DM have focused on reduction of cardiovascular outcomes. These results suggest that intensive treatment does not adversely affect patient-reported outcomes. There have been few cognition studies. Identification of cognitive domains most affected by DM can lead to targeted risk modification, possibly through lifestyle interventions (diet/physical activity) and may reduce risk of cognitive dysfunction and possibly dementia. An overview of cognitive testing in DM showed impairment in tests of executive function, working memory, psychomotor and attentional functions. Impairments of executive function and choice reaction time may have consequences for everyday functioning. Trail Making Task, Symbol Digit Modalities Test, Verbal Fluency Task and tests of reaction time and processing speed could be included as core components of test batteries in future intervention studies.

However there are few studies with a multifactorial intervention and cognition as an endpoint in DM.

FINGER showed that an intensive multi-domain lifestyle intervention programme (nutrition, exercise, cognitive stimulation and social activity, intensive vascular risk factor control) applied in older people (60-77 years) at higher risk for dementia produced significant cognitive benefits after 2 years.

There are concerns whether the intensive nature of the FINGER intervention are translatable/applicable to clinical practice in different healthcare systems. Further studies are required to evaluate the efficacy of multi-domain lifestyle interventions in targeted high-risk populations including a need to develop a practical and feasible program which is deliverable in community settings.

A phase 1 qualitative study (REC ref 19/NI/0011) with our target population generated important data to inform the current study protocol. The theoretical domains framework was used to map the qualitative data, refine implementation approaches and identify active intervention components to support behaviour change. Based on the phase 1 study findings, we have adapted the FINGER multicomponent intervention for use in the context of adults with Type 2 DM in a community setting in Ireland. The study protocol has now been amended to ensure patient and staff safety for delivery of the interventions during the ongoing coronavirus pandemic. We wish to test the acceptability/feasibility of this culturally tailored multicomponent intervention for prevention of cognitive impairment in the target population using a RCT design.

PLAN OF INVESTIGATION Study Design This proposal comprises a 9-month evaluation feasibility/pilot study using parallel group RCT design. Participants will be recruited from both sides of the border using 2 study centres: Sligo (catchment Sligo/Leitrim/West Cavan) and South Western Area Hospital, (SWAH-catchment Tyrone/Fermanagh).

Methodologies

A total of 140 (70 from Sligo/Leitrim/West Cavan and 70 from Tyrone/Fermanagh) non-demented individuals aged ≥ 50 years within 5 years of Type 2 DM diagnosis will be recruited. Those eligible and willing to take part will give informed written consent, and will be randomized to either intensive lifestyle intervention or control (35 participants in each group in each site). All participants will receive general information on brain health in DM at baseline. Participants randomised to control group will receive standard clinical care and be provided with pedometers to wear to record their walking activity while those randomised to the intensive lifestyle intervention will receive a community-based multicomponent programme involving a 4-month active intervention delivered online, followed by a 2-month self-directed consolidation stage. The 4-month active intervention will involve online delivery of the following components:

1. Diet
2. Physical Activity
3. Cognitive stimulation
4. Metabolic and vascular risk factor management.

The 4-month active intervention will be followed by a 2-month self-directed consolidation phase that will include:

* Fortnightly text message reminders as above regarding program targets to include: diet/cognitive stimulation/ exercise/ vascular risk awareness
* Monthly phone calls from the study nurse17 to discuss any issues arising and encourage compliance with the intervention18. The study nurse will telephone participants to review progress in achieving MIND diet and activity and brain training goals and offer positive reinforcement, encouragement and support to continue with the lifestyle changes.
* Participants will also be able to telephone the nurse outside the scheduled calls if and when required.

All participants will then be left to their own initiative for a further 3 months. Participants will meet the researcher at SWAH research centre or their home at baseline, 4, 6 and 9 months for a study assessment that is anticipated to last no longer than 90 minutes. Study visits will be conducted according to local SWAH covid19 protocols and research staff will wear recommended personal protective equipment. Each study visit will involve obtaining a non-fasting blood sample, measurement of blood pressure and anthropometrics (weight, height, waist circumference) and completion of questionnaires. Primary outcomes will include feasibility measures: participation rates; drop-outs; compliance; application of prescribed trial methodology. Acceptability and compliance with these lifestyle interventions will be assessed formally using validated patient questionnaires at each time-point and through interviews with compliers and non-compliers including a sample of participants who dropped out. Secondary outcomes will be global cognitive function, cardiometabolic risk factors and physical performance.

Behavioural measures Diet: Four-day prospective food records, MIND diet score questionnaire. Exercise: muscle strength training and aerobic exercise will be recorded in diaries; participants will be provided with pedometers for objective exercise assessment.

Cognition/social: Activity diaries will quantify participation in social and cognitive activities and use of cognitive training platform (time, frequency and nature of activities). The Brain HQ platform allows recording of the extent of cognitive training.

Health Measures:

Vascular and metabolic risk factors: pulse and blood pressure, glycated haemoglobin (HbA1c), weight, Body Mass Index (BMI), waist circumference, lipid profile, cholesterol, renal function Cognitive and psychological functions will be formally measured using Catch-Cog, Trail Making Test and Delayed Word Recall tests at each assessment.

Physical performance will be measured using 'timed get up and go' and '6-minute walk test' at each assessment.

The need for use of controls This study will test the value of an intensive intervention regimen in people with Type 2 DM. It is important to study acceptability and adherence to such an intervention and to examine whether adherence results in any changes in predefined outcomes, particularly uptake of lifestyle recommendations. Thus, it is necessary to randomly allocate patients with Type 2 DM to a control group to receive routine care. From an ethical perspective the control group will receive the standard of clinical care as defined by national guidelines.

Data protection issues All data will be collected and stored according to Data Protection legislation (NI and ROI). Subjects will be allocated a unique study number so they cannot be identified individually and these databases will be stored separately. Data for this study will be stored securely, according to each institutional data protection policy. For example, within the UK, data is stored according to the Data Protection Act. Similarly, using the UK as an example, stringent internal processes are followed. The Centre for Public Health (CPH) senior management team regularly reviews Quality Control procedures in place within the Centre. CPH have systems in place to ensure that all data handling is carried out in accordance with rigorous internally controlled quality assurance standards with particular attention to confidentiality, data protection and data archiving. Data collected in association with this study will be anonymised and archived in password-protected study databases and will be retained for 10 years in accordance with UK RC policy.

Methods of data collection, and methods of data analysis Baseline assessment, 4 and 6 months assessments: full demographic characteristics {(age, social class and/ or educational attainment) gender, comorbidity, medication, BMI, weight, bloods}); Cognitive and physical performance assessment using Catch Cog, Trails and delayed word recall tests; timed get up and go and six minute walk tests. Primary outcomes include feasibility measures: participation rates; drop-outs; compliance; qualitative (FG) and questionnaire based evaluation of trial processes; application of prescribed trial methodology. Feasibility and compliance with these interventions will also be formally assessed using questionnaires and through Focus Groups, sampling participants to ensure maximum variability and representation of hard to reach groups. Data collection will involve paper methods for all questionnaires and outcomes. Cognitive training records will be obtained from online activity.

Further steps needed and/or envisaged outcome for future work The objective is to proceed to a definitive large-scale study. Our findings will enable refinement of protocol and statistical powering to provide a detailed application to funders for a study that is of high public health priority and that should be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 2 Diabetes mellitus
2. aged ≥50 years
3. within five years of diagnosis
4. access to a computer, tablet or smartphone -

Exclusion Criteria:

1. conditions affecting safe engagement in the intervention (especially the exercise component)
2. insulin therapy
3. malignant diseases
4. major depression within 6 months
5. dementia/substantial cognitive decline
6. Mini Mental State Examination <20
7. symptomatic cardiovascular disease
8. revascularization within 1 year
9. severe loss of vision, hearing, or communicative ability
10. conditions preventing cooperation as judged by the study physician
11. coincident participation in any intervention trial. -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of recruitment strategies, retention, attrition rates and reasons for withdrawal for study participants in both intervention and control groups | at 6 months. T
  This is a feasibility study. we need to collect data on recruitment strategies. We will maintain a record of how many people were contacted, how many consented, the numbers dropping out and the reasons for withdrawal
Determination of fidelity of implementation, feasibility and acceptability of the intervention | at 6 months.
  we will record subject compliance with the study intervention and the feasibility of that intervention. by a questionnaire
Generation of variability data on the primary outcome measure (cognition) from baseline to 6 months on which to base a formal power calculation for a large-scale trial | 6 months.
  Cognition will be assessed using CATCH COG

CONTACTS AND LOCATIONS:
Locations (1):
- South West Acute Hospital, Enniskillen, Co Fermanagh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McEvoy CT, McCarthy G, Townsend RF, Dolan C, Regan-Moriarty J, Cardwell C, McGuinness B, Kennelly SP, Kelly J, McHugh C, Kee F, Bartlett J, Bradshaw C, Reynolds O, Mortland V, O'Neill C, McLoughlin I, McCaffrey N, Heffernan M, Nolan C, Passmore PA. BRAIN-Diabetes: a randomised trial to test the feasibility of an adapted FINGER multidomain intervention in adults with type 2 diabetes living in rural border regions of Ireland. Eur J Ageing. 2025 Jun 24;22(1):30. doi: 10.1007/s10433-025-00862-0. PMID 40550886